CLINICAL TRIAL: NCT04945590
Title: Virtual Intervention and Direct Assessment (VIDA) of Social Determinants of Health in Southern Minnesota Latino Communities After Coronavirus Disease 2019 (COVID-19): a Pilot Study. the VIDA After COVID Study.
Brief Title: The VIDA After COVID Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alice Gallo De Moraes, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-002083
Record Dates: First submitted 2021-06-29; First posted 2021-06-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Latino/Hispanic Virtual Intervention Program (Experimental): Latino/Hispanic individuals will participate in culturally tailored virtual intervention program following a community-based collaborative design.
  Interventions: Behavioral: Virtual Intervention Program

INTERVENTIONS:
Behavioral: Virtual Intervention Program — Four separate virtual individual and group interviews (via telephone or online), which will be scheduled with the help of champions and leaders of the Latino community who will collaborate as companions to improve the commitment and experience of families.

SUMMARY:
The purpose of this study is to objectively identify and address social determinants of health (SDOH) priorities and barriers in Latino patients who survived or are vulnerable to COVID-19, and to understand the consequences of COVID-19 survivorship in local Latino communities.

ELIGIBILITY:
Inclusion Criteria:

* Study population will be identified via community partnerships and peer referrals.
* Participants include Latino families in Southern Minnesota (Dover, Olmsted and Mower county, Minnesota) who survived COVID-19 after requiring ICU or hospital admission, and their families and/or their care partners, or Latino patients who are vulnerable to COVID-19, that have provided research authorization o identified via electronic health registries (following Institutional Review Board approved guidelines).

Exclusion Criteria:

* Families that do not identify as Latino.
* Those living outside Dover, Olmsted and Mower County, Minnesota.
* Those that do not provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Social Determinants of Health (SDOH) Assessment Completed | Through study completion, approximately 3 months
  Number of families in whom SDOH were assessed at baseline and follow-up interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gallo De Moraes, MD, Principal Investigator — Mayo Clinic